CLINICAL TRIAL: NCT01157000
Title: An Open-Label, Single-Dose Study to Assess the Absolute Oral Bioavailability and Pharmacokinetics of JNJ-28431754 (Canagliflozin) Administered as a 300-mg Oral Tablet and an Intravenous Microdose of 10 mcg 14C-canagliflozin in Healthy Male Subjects
Brief Title: A Pharmacokinetic and Bioavailability Study of 28431754 (Canagliflozin) in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CR017197; 28431754DIA1021
Record Dates: First submitted 2010-07-01; First posted 2010-07-05 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Healthy
Keywords: Canagliflozin; Pharmacokinetic; Bioavailability
MeSH Terms: interventions — Canagliflozin

ARMS (1):
- 001 (Experimental): Canagliflozin On Day 1 all patients will receive a single 300-mg tablet of canagliflozin with 8 ounces of water followed 105 minutes later by a 15-minute intravenous infusion dose (15 mL) of 10 mcg of 14C-canagliflozin (200 nCi).
  Interventions: Drug: Canagliflozin

INTERVENTIONS:
Drug: Canagliflozin — On Day 1, all patients will receive a single 300-mg tablet of canagliflozin with 8 ounces of water followed 105 minutes later by a 15-minute intravenous infusion dose (15 mL) of 10 mcg of 14C-canagliflozin (200 nCi).

SUMMARY:
The purpose of this study is to evaluate the absolute oral bioavailability (how fast and how much study drug is absorbed in the body) of a single 300-mg oral dose of canagliflozin in healthy male volunteers.

DETAILED DESCRIPTION:
This is an open-label (the patient will know the identity of the treatment they receive), single-dose, single-center study to evaluate the absolute oral bioavailability (the rate and extent at which the drug is absorbed in the body and reaches blood circulation) of a 300-mg tablet of canagliflozin. Approximately 9 healthy men (referred to as healthy male volunteers) will receive a single 300-mg tablet of canagliflozin with an 8 ounce glass of water followed 105 minutes later by a 15 minute intravenous (iv) infusion (administration directly in the vein) of a very small dose (ie, 10 micrograms [mcg]) of canagliflozin that has been combined with a radioactive carbon isotope referred to as 14C canagliflozin. The radiolabelled 10 mcg dose of canagliflozin will act as a tracer to measure the total amount of canagliflozin that is absorbed and metabolized in the body. After dosing, blood, urine and feces samples will be collected for pharmacokinetic and safety evaluations at specified timepoints for up to 72 hours. The primary outcome measure in the study is to determine the absolute bioavailability of a single 300 mg dose of canagliflozin by estimation of protocol-specified standard plasma pharmacokinetic parameters (parameters that measure the absorption, distribution, metabolism, and elimination of drug by the body) from blood samples obtained during the study. During the study, the safety of a single oral 300-mg dose of canagliflozin administered together with a single iv 10-mcg infusion dose of 14C-canagliflozin will be evaluated by monitoring adverse events and findings from clinical laboratory test values, physical examination results, 12 lead ECGs and vital signs measurements reported. On Day 1, each healthy volunteer will take a single 300-mg canagliflozin tablet orally (by mouth) with 8 ounces of water in the morning followed by a 15-minute intravenous infusion of 10 mcg 14C-canagliflozin (200 nCi) (equivalent to 0.666 mcg/mL of canagliflozin). Healthy volunteers will fast at least 10 hours before dosing and until at least 4 hours after oral administration and will not be allowed to drink water from 2 hours before and up to 4 hours after study drug administration.

ELIGIBILITY:
Inclusion Criteria:

* Signed an informed consent document indicating they understand the purpose of and procedures required for the study and are willing to participate in the study
* agrees to use an adequate contraception method as deemed appropriate by the investigator (e.g., vasectomy, double-barrier, partner using effective contraception) and to not donate sperm during the study and for 3 months after receiving the last dose of study drug
* has a blood pressure (after sitting for 5 minutes) between 90 and 140 mmHg systolic, inclusive, and no higher than 90 mmHg diastolic

Exclusion Criteria:

* Used any 14C labeled medication within 6 months before the first dose of the study drug is scheduled
* Have history of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the subject or that could interfere with the interpretation of the study results
* Have clinically significant abnormal values for hematology, clinical chemistry or urinalysis at screening and at admission to the study center as deemed appropriate by the investigator
* Have clinically significant abnormal physical examination, vital signs or 12 lead ECG at screening and admission to the study center as deemed appropriate by the investigator
* Used any prescription or nonprescription medication (including vitamins and herbal supplements), except for occasional use of paracetamol (a maximum of 3 doses per day of 500 mg paracetamol, and no more than 3 grams per week), within 14 days before the first dose of the study drug is scheduled

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2010-05; Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Protocol-specified pharmacokinetic parameters from blood samples to assess the absolute bioavailabilty of a 300-mg oral dose of canagliflozin | Predose on Day 1 up to 72 hours postdose

SECONDARY OUTCOMES:
Protocol-specified pharmacokinetic parameters from blood samples to evaluate the pharmacokinetics of a single 300-mg oral dose of canagliflozin administered with a single 10-mcg intravenous dose of 14C canagliflozin | Predose on Day 1 up to 72 hours postdose
Measurement of 14C radioactivity from total urine and feces output to evaluate the extent of biliary excretion of a single 10-mcg intravenous dose of 14C canagliflozin | Day 1 through 72 hours after initiation of the intravenous infusion
The number and type of adverse events reported | Time of screening up to 5 to 7 days after completion of all study related procedures on Day 4

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Merksem, Belgium

REFERENCES:
- [Derived] Devineni D, Murphy J, Wang SS, Stieltjes H, Rothenberg P, Scheers E, Mamidi RN. Absolute oral bioavailability and pharmacokinetics of canagliflozin: A microdose study in healthy participants. Clin Pharmacol Drug Dev. 2015 Jul;4(4):295-304. doi: 10.1002/cpdd.162. Epub 2014 Dec 11. PMID 27136910